| GCS Co., Ltd. | GANA V <sup>®</sup> | Final version 5.0 | Confidential |
|---------------|---------------------|-------------------|--------------|
| | CIP #21E0787 | Date: 27/06/2022 | Page 1/6 |

## OVERALL SYNOPSIS OF THE CLINICAL INVESTIGATION # 21E0787

| ANSM registration #: | 2021-A02451-40 |
|---|---|
| Clinical investigation plan #: | 21E0787 |
| Title of the clinical investigation: | Clinical study for the safety and effectiveness of use of an injectable medical device GANA V <sup>®</sup> for facial aesthetic treatment |
| Sponsor: | GCS Co., Ltd. 1008 Ho, Sunil Technopia Bldg, 555 Dunchon-daero Jungwon-gu, Seongnam-si, Gyeonggi-do KOREA |
| Development phase | Post market study Interventional Device used according to Instruction For Use (IFU) |
| Objectives: | The primary objective is to evaluate the effectiveness of Gana V® in comparison with Sculptra® in the correction of Nasolabial Folds (NLFs) 6 months after treatment initiation. The secondary objectives of the study are: - To evaluate the effectiveness of Gana V® in comparison with Sculptra® in the correction of Nasolabial Folds (NLFs) 1¹¹², 3, 9, 12, 18 and 24 months after treatment initiation. - To evaluate the effectiveness of Gana V® in comparison with Sculptra® on the global aesthetic improvement 1¹¹², 3, 6, 9, 12, 18 and 24 months after treatment initiation. - To evaluate the effectiveness of Gana V® in comparison with Sculptra® in reducing NLFs depth and volume 1¹¹², 3, 6, 9, 12, 18 and 24 months after treatment initiation. - To evaluate the subject satisfaction with Gana V® in comparison with Sculptra® 1¹¹², 3, 6, 9, 12, 18 and 24 months after treatment initiation. - To evaluate the injector satisfaction with Gana V® in comparison with Sculptra® after initial injection and touch-up injection if applicable. - To evaluate the safety of Gana V® in comparison with Sculptra®. |
| Design: | The study will be: |
| Planned Sample Size: | 55 subjects randomized. |
| Number of investigational study sites: | 1 site (France) |
| Inclusion criteria: | <ol> <li>Healthy Subject</li> <li>Sex: male or female</li> <li>Age: between 30 and 70 years.</li> <li>Subject with moderate to severe nasolabial folds as determined by a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 on both folds at the pre-treatment evaluation.</li> </ol> |

| GCS Co., Ltd. | GANA V <sup>®</sup><br>CIP #21E0787 | Final version 5.0<br>Date: 27/06/2022 | Confidential<br>Page 2/6 |
|---|---|---|---|
| | fillers, to peels, n period. 6. Subject, information consent. 8. Subject v. 9. Subject a 10. Female regimen | xin treatments, laser, micron-invasive skin-tightening psychologically able to uron and to give a written information properties and willing to have photographs affiliated to a health social sof childbearing potential second control of the se | expressly his/her informed of the face taken. ecurity system. should use a contraceptive ce at least 12 weeks before |
| Exclusion criteria: | study. 2. Subject of the face | rative or legal decision or we had social or sanitary estable participation to another research exclusion period of one having received 4500 cion in research involving months, including participal suspected to be non-contor's judgment. Suffering from a severe or pathology that may interfere sults. With known history of or seand/or immune deficiency, suffering from inflamments disorders in or near the papilloma, chronic eczes with labial herpes in the last omatic at time of screening with an abscess, unhealed brous lesion on the studied approne to develop inflamment of the test of the test having history of allergy the components of the test having received treatments on the face withing the face area within the green the face area within the green the second of the test of | at disorders or anything on the evaluation. The evaluation of their freedom by the is under guardianship. The earch on human beings or euros indemnities for human beings in the 12 tion in the present study. The evaluation of the |

| GCS Co., Ltd. | GANA V <sup>®</sup><br>CIP #21E0787 | Final version 5.0<br>Date: 27/06/2022 | Confidential<br>Page 3/6 |
|---|---|---|---|
| | filling primethacry the face. 18. Subject If threads of the subject hor visit. 20. Subject inflamma antiplatel prolong because a systemic • Antifi • Immurprior • Retir 22. Intensive | <ol> <li>Subject having received at any time a treatment with tensor threads on the face.</li> <li>Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit.</li> <li>Subject using medication such as aspirin, nonsteroidal anti inflammatory drugs (NSAID) (ibuprofen, naproxen,) antiplatelet agents, anticoagulants or other substances known to prolong bleeding time within 1 week prior to injection visits.</li> <li>Subject undergoing a topical treatment on the test area or a systemic treatment: <ul> <li>Antihistamines during the 2 weeks prior to screening visit.</li> </ul> </li> </ol> | |
| Investigational device Name / code Classification Composition Galenic form Administration route | Gana V® Class III med Poly-L-Lactic Mannitol. Sterile freeze | ical device | Carboxymethyl Cellulose, |
| Comparator: Name / code Classification Composition Galenic form Administration route | Sculptra® Class III med Poly-L-Lactic Mannitol. Sterile freeze | ical device | Carboxymethyl Cellulose, |
| Endpoints: | Primary effect Mean change treatment initial evaluator usit (WSRS). Secondary effect - Mean change treatment initial evaluator usit (WSRS). Secondary effect in Mean 24 mm live in 10 | e in NLFs severity from tiation, as assessed by any the validated 5-point Wrong the valuator. The valuator of the | baseline to 6 months after an independent blinded live rinkles Severity Rating Scale eline to 11/2, 3, 9, 12, 18 and ion as assessed by a blinded 6, 9, 12, 18 and 24 months assessed by a blinded live inder is defined as a subject ment from baseline on the occale (GAIS) responder rates after treatment initiation a blinded live independent fined as a subject having |

| GCS Co., Ltd. | GANA V <sup>®</sup><br>CIP #21E0787 | Final version 5.0<br>Date: 27/06/2022 | Confidential<br>Page 4/6 |
|---|---|---|---|
| | acco<br>- Mea<br>3, 6,<br>fring<br>- Prop<br>mon<br>- Inject<br>and | ording to GAIS. In change in NLF depth and 9, 12, 18 and 24 months a e projection system. In ortion of satisfied subjects ths after treatment initiation | injection quality after initial |
| | Investigation<br>Injection Site | al devices safety will be<br>Reactions (ISRs) and Adve<br>the investigator. Subjects | assessed by collection of<br>erse Events (AEs) throughout<br>will record ISRs and AEs in |
| Study Procedures: | A screening | A screening visit will allow to inform and preselect the subjects. | |
| | photographs<br>receive a firs<br>randomizatio<br>satisfaction<br>Adverse Ev | will be done before injet injection of the investigation list. Immediately after in will be collected. Investigation | e projection acquisitions and ction. Eligible subjects will onal devices according to the njection, injector's treatment gator evaluator will collect on Site Reactions (ISRs) |
| | scoring, fring<br>before touch<br>injector's tre<br>touch-up inje<br>subject opin | e projection acquisitions and up (if applicable). Subject atment satisfaction (if appliction will be made if necess | n (M1 <sup>1/2</sup> ), WSRS and GAIS<br>nd photographs will be done<br>is treatment satisfaction and<br>licable) will be collected. A<br>ary, according to injector and<br>will collect AEs and ISRs |
| | twenty-four (<br>(WSRS and<br>photographs | Three (M3), six (M6), nine (M9), twelve (M12), eighteen (M18) and twenty-four (M24) months after initial injection, effectiveness scoring (WSRS and GAIS scales), fringe projection acquisitions and photographs will be done. Subject's treatment satisfaction will be collected. Investigator evaluator will collect AEs and ISRs | |
| Statistical methods: | For the prim | nary evaluation criterion: | |
| | level scores (<br>statistics for<br>deviation, firs | (at D0 before injection and N<br>quantitative variable (N<br>st and third quartile, minim | g Scale (WSRS) with the <u>5</u> /16) will be summarized using, mean, median, standard um and maximum value) for ge from baseline (M6-D0bef) |
| | Inferential a | nalysis for the primary er | ndpoint: |
| | if the upper- | | culptra <sup>®</sup> will be demonstrated<br>CI of the (M6-D0bef) mean |
| | For the second | For the secondary evaluation criteria: | |
| | to their type (<br>For quantitat | All the variables will be described using adapted statistics according to their type (quantitative data or qualitative data). For quantitative data a Wilcoxon or paired t test will be applied assess the change from baseline and to compare the products. | |

| GCS Co., Ltd. | GANA V <sup>®</sup> | Final version 5.0 | Confidential |
|---------------|---------------------|-------------------|--------------|
| | CIP #21E0787 | Date: 27/06/2022 | Page 5/6 |

| | For qualitative data a McNemar's test will be applied to compare the proportion of improvement or satisfaction between the products. |
|---|---|
| | The bilateral approach will be used with a significance level of 0.05. |
| Foreseen study duration: | Clinical investigation beginning: Q1 2022 |
| | Clinical investigation end: Q2 2024 |
| | Clinical investigation global duration: 28 months |
| | Duration by subject: 24 months + screening period |

| GCS Co., Ltd. GANA V® Final version 5.0 Confidential CIP #21E0787 Date: 27/06/2022 Page 6/6 |
|---|
|---|

## FLOW-CHART

| | FLOW-CHART | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | Visit 1<br>Screenin<br>g | Visit 2<br>Day 0 | Visit 3<br>M1 <sup>1/2</sup> | Visit 4<br>M3 | Visit 5<br>M6 | Visit 6<br>M9 | Visit 7<br>M12 | Visit 8<br>M18 | Visit 9<br>M24 |
| Days | D-x | D0 | D40<br>±2 | D90<br>±2 | D180<br>±4 | D270<br>±4 | D365<br>±7 | D540<br>±14 | D730<br>±14 |
| Informed consent form signature | • | | | | | | | | |
| Medical examination | • | | | | | | | | |
| Medical history and previous and concomitant treatments collection | • | | | | | | | | |
| Checking of the inclusion and exclusion criteria | • | | | | | | | | |
| Pregnancy test | | ●b | | | | | | | |
| Confirmation of eligibility | | ●b | | | | | | | |
| Randomization | | • | | | | | | | |
| WSRS live assessment by a blinded evaluator | • | ●p | <b>●</b> b | • | • | • | • | • | • |
| Macrophotographs | | ●b | ●p | • | • | • | • | • | • |
| Fringe projection acquisitions (2 areas) | | <b>●</b> b | <b>●</b> b | • | • | • | • | • | • |
| Injection + anaesthesia (if necessary) | | • | ●Touch up | | | | | | |
| GAIS live assessment by a blinded evaluator | | | <b>●</b> b | • | • | • | • | • | • |
| GAIS assessment by the subjects | | | <b>●</b> b | • | • | • | • | • | • |
| Subjective evaluation questionnaire for subjects | | | <b>●</b> b | • | • | • | • | • | • |
| ISR assessor | | ●a | ●b + a | • | • | • | • | • | • |
| ISR subjects | | completed each day during 4 weeks after injection and touch up if applicable at home by the subject | | | | | | | |
| Subjective evaluation questionnaire for injector | | <b>⊕</b> a | ●a | | | | | | |
| AE and concomitant treatments and procedures collection | • | • | • | • | • | • | • | • | • |
| Study end | | | | | | | | | • |

Keys:b: Before injection; a: After injection